CLINICAL TRIAL: NCT05327920
Title: Impact of UPaDacitinib Treatment on inflAmmaTion, AchiEvement of Treatment Targets and Health-related Quality of Life, Work Ability and Healthcare Resource Utilization in Moderate to Severe Rheumatoid Arthritis Patients in Hungarian Real-world Practice
Brief Title: An Observational Study to Assess the Impact of Upadacitinib in Adult Hungarian Participants With Moderate to Severe Rheumatoid Arthritis (RA) in Real-World Practice
Acronym: UPDATE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-125
Record Dates: First submitted 2022-04-12; First posted 2022-04-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis (RA); Upadacitinib; RINVOQ
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for Rheumatoid Arthritis

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. Despite the range of treatment options for RA steadily increasing, many patients remain sub-optimally managed, with sustained clinical remission rarely achieved. This study will assess the impact of upadacitinib treatment on achievement of remission and low disease activity in moderate to severe RA Hungarian patients in the real-world setting.

Upadacitinib is an approved drug for the treatment of adults with moderately to severely active RA. Adult participants with moderate-to-severe RA will be enrolled. Around 90 participants who are prescribed upadacitinib in routine clinical practice will be enrolled in the study in approximately 8 sites in Hungary.

Participants will receive upadacitinib as prescribed by the physician and will be followed for approximately 12 months.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic and only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe active rheumatoid arthritis (RA) upon judgment of the treating physician.
* Upadacitinib prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies and upadacitinib treatment was started within 1 week before the enrollment.
* Physician decision on participant treatment with upadacitinib must have been reached prior to and independently of recruitment in the study.

Exclusion Criteria:

* Participants who cannot be treated with upadacitinib as per SmPC or local prescription criteria.
* Prior treatment course with upadacitinib or the current upadacitinib treatment was started more than 1 week prior to enrollment.
* Participant currently participating in any interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Participants with moderate-to-severe rheumatoid arthritis (RA).
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving 28-Joint Disease Activity Score (DAS28) C-reactive protein (CRP) Remission following initiation of treatment with Upadacitinib | 6 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Remission is defined as a DAS28 CRP <2.6.

SECONDARY OUTCOMES:
Percentage of Participants Achieving DAS28 CRP Remission following Initiation of Treatment with Upadacitinib | Up to 12 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Remission is defined as a DAS28 CRP <2.6.
Percentage of Participants Achieving DAS28 CRP Remission at month 6 and maintain it in all subsequent visits | Up to 12 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Remission is defined as a DAS28 CRP <2.6.
Percentage of Participants Achieving DAS28 CRP Low Disease Activity (LDA) following Initiation of Treatment with Upadacitinib | Up to 12 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Low disease activity is defined as DAS28 CRP <=3.2.
Percentage of Participants Achieving DAS28 CRP Low Disease Activity at month 6 and maintain it in all subsequent visits | Up to 12 Months
  The DAS28 CRP is a composite measure of a patient's level of disease activity at a given time. The score ranges from 0-9.4 with a higher score correlating to higher disease activity. Low disease activity is defined as DAS28 CRP <=3.2.
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score | Up to 12 Months
  The HAQ-DI assesses physical function in RA. The HAQ-DI score is the average of the highest score in each of eight categories. The total score is between 0-3.0, in 0.125 increments. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment
Change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score | Up to 12 Months
  The FACIT-Fatigue Scale measures an individual's level of fatigue during their usual daily activities over the past week on a four-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The score range for FACIT-Fatigue is between 0 and 52. A score of less than 30 indicates severe fatigue. The higher the score, the better the quality of life.
Change from Baseline in EQ-5D-5L Score | Up to 12 Months
  The EQ-5D-5L comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The respondent selects one of three different levels of problem severity. The levels are none, moderate and severe/extreme (coded 1 through 3, respectively).
Change from Baseline in Morning Stiffness Visual Analogue Scale (VAS) Score | Up to 12 months
  The participant's level of morning stiffness in the past 7 days will be measured using a VAS. VAS scores range from 0 to 100 points with a higher score indicating severity of morning stiffness.
Change from Baseline in the Treatment Satisfaction Questionnaire for Medication (TSQM) Score | Up to 12 Months
  TSQM scores have a range of 0 to 100, with higher scores indicating higher satisfaction. The 14 items of the TSQM cover four domains: Effectiveness, Side Effects, Convenience, and Global Satisfaction.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire-Rheumatoid Arthritis (WPAI-RA) Score | Up to 12 Months
  The WPAI-RA measures the impact of health problems on presenteeism, absenteeism, total work productivity impairment, total activity impairment using a 0 to 10 VAS.
Health Resource Utilization (HRU) Questionnaire - Difference in the Number of Hospital Inpatient Days | 12 months prior to month 0 (baseline) and 12 months prior to month 12
  Difference in the number of hospital inpatient days during 12 months of upadacitinib therapy and 12 months preceding the introduction of upadacitinib therapy.
HRU Questionnaire - Difference in the Number of Hospitalizations | 12 months prior to month 0 (baseline) and 12 months prior to month 12
  Difference in the number of hospital inpatient days during 12 months of upadacitinib therapy and 12 months preceding the introduction of upadacitinib therapy.
HRU Questionnaire - Difference in the Number of Sick Leave Days (in employed subjects only) | 12 months prior to month 0 (baseline) and 12 months prior to month 12
  Difference in the number of hospital inpatient days during 12 months of upadacitinib therapy and 12 months preceding the introduction of upadacitinib therapy.
HRU Questionnaire - Difference in the Number of Sick Leaves (in employed subjects only) | 12 months prior to month 0 (baseline) and 12 months prior to month 12
  Difference in the number of sick leaves during 12 months of upadacitinib therapy and 12 months preceding the introduction of upadacitinib therapy.
HRU Questionnaire - Difference in the Number of Outpatient Visits to Each Kind of Health Care Provider | 12 months prior to month 0 (baseline) and 12 months prior to month 12
  Difference in the number of outpatient visits to each kind of health care provider which includes general practitioner, rheumatologist, other specialists (ophthalmologist, gastroenterologist, dermatologist, physiatrist), physiotherapist and rheumatology nurses during 12 months of upadacitinib therapy and 12 months preceding the introduction of upadacitinib therapy.
Percentage of Participants remaining on Upadacitinib treatment | Up to 12 Months
  Percentage of participants remaining on upadacitinib up to 12 months post initiation.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- Hungary (8):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 234201, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem-Klinikai Kozpont /ID# 246156, Debrecen, Hajdú-Bihar
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 234204, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz /ID# 239231, Gyula
  - Kistarcsai Flor Ferenc Korhaz /ID# 234202, Kistarcsa
  - BAZ Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz /ID# 246158, Miskolc
  - Szegedi Tudományegyetem /ID# 244364, Szeged
  - MÁV Kórház /ID# 246157, Szolnok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P22-125#additional-resources-section